CLINICAL TRIAL: NCT04416256
Title: Consequences of the COVID-19 Pandemic on Worldwide Organ Procurement and Transplantation
Brief Title: COVID-19 Pandemic and Worldwide Organ Procurement
Acronym: COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Collaborators: Agence de La Biomédecine (Other Government); Eurotransplant (Unknown); United Network for Organ Sharing (Unknown); Deutsche Stiftung Organtransplantation (Unknown); Centro Nazionale Trapianti (Unknown); Brazilian Organ Transplant Association (Unknown); The Canadian Association of Transplantation (Unknown); Scandiatransplant (Unknown); Nederlandse Transplantatie Vereniging (Unknown); Austrotransplant (Unknown); Centro Nacional de Trasplantes (Unknown); Instituto Nacional de Donación y Trasplante de Células, Tejidos y Órganos (Unknown); Donor Network of Croatia (Unknown); Instituto Nacional Central Único Coordinador de Ablación e Implante (Other Government); Corporación Nacional de Trasplantes de Chile (Unknown); Australian Organ and Tissue Donation and Transplantation Authority (Unknown); Organización Nacional de Trasplantes (Unknown); Autoridade Para Services de Sangue e Transplantacáo (Unknown)
Responsible Party: Sponsor
Other Study IDs: COVID/W.W.
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: organ; procurement; transplantation; pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (18):
- France: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Spain: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Portugal: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Croatia: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Germany: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Italy: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Netherlands: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Austria: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- US: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Canada: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Mexico: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Brazil: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Uruguay: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Argentina: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Chile: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Australia: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Belgium: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.
- Finland: All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.

SUMMARY:
End-stage organ failure is estimated to affect more than 4 to 6 million persons worldwide. In 2018, transplant systems across the globe enabled around 150,000 patients to benefit from a kidney, heart, lung, liver, or other solid organ, a number that was far less than the demand. According to data from the World Health Organization, more than 1,500,000 persons live with a transplanted organ worldwide. In the US, approximately 40,000 patients receive an organ transplant every year, but 120,000 still remain waitlisted for transplantation today, with 7,600 dying annually while waiting for an organ transplant. A similar lack of organs and high death rates on the waiting list affect patients in Europe and many other countries.

As nations adjust to new realities driven by the coronavirus (COVID-19) outbreak, many health care providers, institutions and patients are concerned about the potential impact that COVID-19 will have on organ donation and transplantation. One concern is that transplant recipients may have a greater susceptibility to infection and greater viral burden. A second concern is that hospitals will lack the resources in terms of staff and equipment to care for recipients after transplantation, who often require intensive care and multispecialty management.

Because of the overwhelming healthcare system burden, a dramatic negative effect on worldwide organ donation and transplantation is anticipated, but has not been measured. Our objective was to quantify the worldwide impact of COVID-19 pandemic on organ donation and transplantation and consequences for waitlisted patients.

ELIGIBILITY:
Inclusion Criteria:

* All organs procured for transplantation and transplanted during the observation period. These include kidney, lung, liver, heart, and combined transplantations.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Solid organ transplants performed during the study period (kidney, lung, heart, liver and combined organs in Europe (France, Spain, Portugal, Germany, Italy, Croatia, Belgium, Netherlands, Austria), North America (US and Canada), Central and South America (Mexico, Brazil, Uruguay, Argentina and Chile) and Oceania (Australia)
Sampling Method: Non-Probability Sample
Enrollment: 230000 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Organ transplantation activity during COVID-19 pandemic | Two years since COVID-19 outbreak.
  Overall deceased donor transplantation performed during the COVID-19 pandemic. Stratified analysis by deceased donor type (Kidney, lung, Liver, heart), and combined transplantations during the COVID-19 pandemic.

SECONDARY OUTCOMES:
Further analysis on organ transplantation with stratification | Two years since COVID-19 outbreak.
  Geographic disparities related to organ transplantation rates and association with COVID-19 clusters Living donor transplantation performed during the COVID-19 pandemic. Quality of transplanted organs (kidney) before and after the COVID-19 pandemic. Change in relationship between living donors and their recipients before and after the COVID-19 pandemic.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, Principal Investigator — Paris Translational Research Center for Organ Transplantation
Locations (1):
- Paris Transplant Group, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu B, Kraemer MUG; Open COVID-19 Data Curation Group. Open access epidemiological data from the COVID-19 outbreak. Lancet Infect Dis. 2020 May;20(5):534. doi: 10.1016/S1473-3099(20)30119-5. Epub 2020 Feb 19. No abstract available. PMID 32087115
- [Background] Anderson RM, Heesterbeek H, Klinkenberg D, Hollingsworth TD. How will country-based mitigation measures influence the course of the COVID-19 epidemic? Lancet. 2020 Mar 21;395(10228):931-934. doi: 10.1016/S0140-6736(20)30567-5. Epub 2020 Mar 9. No abstract available. PMID 32164834
- [Background] Ahn C, Amer H, Anglicheau D, Ascher NL, Baan CC, Battsetset G, Bat-Ireedui B, Berney T, Betjes MGH, Bichu S, Birn H, Brennan D, Bromberg J, Caillard S, Cannon RM, Cantarovich M, Chan A, Chen ZS, Chapman JR, Cole EH, Cross N, Durand F, Egawa H, Emond JC, Farrero M, Friend PJ, Geissler EK, Ha J, Haberal MA, Henderson ML, Hesselink DA, Humar A, Jassem W, Jeong JC, Kaplan B, Kee T, Kim SJ, Kumar D, Legendre CM, Man K, Moulin B, Muller E, Munkhbat R, Od-Erdene L, Perrin P, Rela M, Tanabe K, Tedesco Silva H, Tinckam KT, Tullius SG, Wong G. Global Transplantation COVID Report March 2020. Transplantation. 2020 Oct;104(10):1974-1983. doi: 10.1097/TP.0000000000003258. No abstract available. PMID 32243281
- [Background] Zhang X. Epidemiology of Covid-19. N Engl J Med. 2020 May 7;382(19):1869. doi: 10.1056/NEJMc2005157. Epub 2020 Mar 27. No abstract available. PMID 32220200
- [Background] Martino F, Plebani M, Ronco C. Kidney transplant programmes during the COVID-19 pandemic. Lancet Respir Med. 2020 May;8(5):e39. doi: 10.1016/S2213-2600(20)30182-X. Epub 2020 Apr 16. No abstract available. PMID 32305079
- [Background] Akalin E, Azzi Y, Bartash R, Seethamraju H, Parides M, Hemmige V, Ross M, Forest S, Goldstein YD, Ajaimy M, Liriano-Ward L, Pynadath C, Loarte-Campos P, Nandigam PB, Graham J, Le M, Rocca J, Kinkhabwala M. Covid-19 and Kidney Transplantation. N Engl J Med. 2020 Jun 18;382(25):2475-2477. doi: 10.1056/NEJMc2011117. Epub 2020 Apr 24. No abstract available. PMID 32329975
- [Background] Coates PT, Wong G, Drueke T, Rovin B, Ronco P; Associate Editors, for the Entire Editorial Team. Early experience with COVID-19 in kidney transplantation. Kidney Int. 2020 Jun;97(6):1074-1075. doi: 10.1016/j.kint.2020.04.001. Epub 2020 Apr 9. No abstract available. PMID 32354635
- [Background] Livingston E, Bucher K. Coronavirus Disease 2019 (COVID-19) in Italy. JAMA. 2020 Apr 14;323(14):1335. doi: 10.1001/jama.2020.4344. No abstract available. PMID 32181795
- [Background] Omer SB, Malani P, Del Rio C. The COVID-19 Pandemic in the US: A Clinical Update. JAMA. 2020 May 12;323(18):1767-1768. doi: 10.1001/jama.2020.5788. No abstract available. PMID 32250388
- [Background] Dong E, Du H, Gardner L. An interactive web-based dashboard to track COVID-19 in real time. Lancet Infect Dis. 2020 May;20(5):533-534. doi: 10.1016/S1473-3099(20)30120-1. Epub 2020 Feb 19. No abstract available. PMID 32087114
- [Result] Levin A, Tonelli M, Bonventre J, Coresh J, Donner JA, Fogo AB, Fox CS, Gansevoort RT, Heerspink HJL, Jardine M, Kasiske B, Kottgen A, Kretzler M, Levey AS, Luyckx VA, Mehta R, Moe O, Obrador G, Pannu N, Parikh CR, Perkovic V, Pollock C, Stenvinkel P, Tuttle KR, Wheeler DC, Eckardt KU; ISN Global Kidney Health Summit participants. Global kidney health 2017 and beyond: a roadmap for closing gaps in care, research, and policy. Lancet. 2017 Oct 21;390(10105):1888-1917. doi: 10.1016/S0140-6736(17)30788-2. Epub 2017 Apr 20. PMID 28434650
- [Derived] Aubert O, Yoo D, Zielinski D, Cozzi E, Cardillo M, Durr M, Dominguez-Gil B, Coll E, Da Silva MI, Sallinen V, Lemstrom K, Midtvedt K, Ulloa C, Immer F, Weissenbacher A, Vallant N, Basic-Jukic N, Tanabe K, Papatheodoridis G, Menoudakou G, Torres M, Soratti C, Hansen Krogh D, Lefaucheur C, Ferreira G, Silva HT Jr, Hartell D, Forsythe J, Mumford L, Reese PP, Kerbaul F, Jacquelinet C, Vogelaar S, Papalois V, Loupy A. COVID-19 pandemic and worldwide organ transplantation: a population-based study. Lancet Public Health. 2021 Oct;6(10):e709-e719. doi: 10.1016/S2468-2667(21)00200-0. Epub 2021 Aug 30. PMID 34474014